CLINICAL TRIAL: NCT01244464
Title: Safety Study of IMOVAX Polio™ in Selected Cities in China, an Observational Post Marketing Study
Brief Title: A Study of the Safety of IMOVAX Polio™ in China
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IPV29; UTN: U1111-1114-3719 (Other: WHO)
Record Dates: First submitted 2010-11-17; First posted 2010-11-19 (Estimated); Last update posted 2012-08-03 (Estimated); Status verified 2012-08

CONDITIONS: Poliomyelitis; Polio
Keywords: Poliomyelitis; IMOVAX POLIO™; Polio
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Group (Experimental)
  Interventions: Biological: IMOVAX Polio™-Inactivated types 1, 2, and 3 poliovirus D vaccine

INTERVENTIONS:
Biological: IMOVAX Polio™-Inactivated types 1, 2, and 3 poliovirus D vaccine — 0.5 mL, at 2, 3, and 4 months; Intramuscular
  Other Names: IMOVAX POLIO™

SUMMARY:
This study is designed to obtain post-marketing safety data on IMOVAX Polio™ vaccine in China.

Primary Objective: To describe the safety profile after each dose of IMOVAX Polio™ administered at 2, 3, and 4 months of age in population aged over 2 months old living in the study city China.

DETAILED DESCRIPTION:
Study participants will receive a single dose of IMOVAX Polio™ vaccine at 2, 3, and 4 months of age, respectively. Each participant will make a total of 7 visits. Safety will be monitored at each visit and up to 30 days after each vaccination.

ELIGIBILITY:
Inclusion Criteria :

* Subject is more than 2 months (60-89 days) old when receiving the first dose of polio vaccine.
* Subject's parents/legal representative showed willingness to complete the 3 primary doses fully using IMOVAX Polio™ according to the schedule: one injection at 2, 3, 4 months old, respectively.
* Informed consent form obtained from the subject's parent/legal representative.
* Subject plan to live in the selected study sites for at least three months after inclusion.

Exclusion Criteria :

* Subject with a history of serious illness (e.g., hypersensitivity, seizure, convulsion, encephalopathy diseases)
* Known or suspected impairment of immunologic function
* Acute medical illness with or without fever within the last 72 hours
* Subject plan to leave the study sites for at least three months after inclusion
* Administration of immune globulin or other blood products within the last three months
* Participation in another clinical trial at the same time
* Contraindication to vaccination according to IMOVAX Polio™ leaflet.

Ages: 60 Days to 89 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 800 (Actual)
Dates: Start 2010-11; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The occurrence, duration, and relationship to vaccination of solicited and unsolicited (spontaneously reported) adverse events occurring after IMOVAX Polio™ vaccination. | Day 0 to Day 30 post-vaccination
  Solicited injection site reactions: tenderness, erythema, and swelling. Solicited systemic reactions: Fever (temperature), vomiting, abnormal crying, drowsiness, loss of appetite, and irritability.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur China
Locations (1):
- Shanghai, China

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com